CLINICAL TRIAL: NCT03118596
Title: Fibre-optic Guided Tracheal Intubation Through Supraglottic Airway Devices - a Randomised Comparison Between I-gel and the LMA ProtectorTM
Brief Title: Fibre-optic Guided Tracheal Intubation Through SADs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHCoventryNHS
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Intubation; Difficult or Failed; Laryngeal Masks; Airway Management
Keywords: intubation; tracheal; airway device; supra-glottic airway device; fibreoptic scope

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-gel (Active Comparator): Fibreoptic guided tracheal intubation through I-gel
  Interventions: Device: I-gel
- LMA Protector (Active Comparator): Fibreoptic guided tracheal intubation through Protector
  Interventions: Device: LMA Protector

INTERVENTIONS:
Device: I-gel — Fibreoptic guided tracheal intubation is going to be performed through the I-gel supraglottic airway.
  Arms: I-gel
Device: LMA Protector — Fibreoptic guided tracheal intubation is going to be performed through the LMA Protector supraglottic airway.
  Arms: LMA Protector

SUMMARY:
The study aims to establish which of the two second generation Supraglottic Airway Devices, the I-gel or the the laryngeal ask airway (LMA) Protector, is best suited to be used as a conduit to fibreoptic bronchoscope assisted tracheal intubation. The primary outcome of this will be the time to complete the tracheal intubation.

DETAILED DESCRIPTION:
Tracheal intubation through a supraglottic airway device (SAD) is a well-established technique in the management of patients with a difficult airway. The technique can be used in patients in whom difficult intubation is expected, or in situations when tracheal intubation using another method was not possible. It is now recommended that tracheal intubation through the SAD should be performed using a fibreoptic scope (a camera device) to minimise the risk of trauma to the airway, and that second generation SADs are used to minimise the risk of aspiration of gastric contents.

There are two second generation SADs currently available which allow tracheal intubation: the I-gel and the LMA protector.

The I-gel is a second generation supraglottic airway device widely used in anaesthesia and resuscitation. Fibreoptic intubation through the I-gel has been evaluated in a recent prospective study (1), with the first attempt success rate of 91.4%. In another study (2) of patients with predicted difficult airway, the success rate of the procedure at first attempt was 96%.

LMA Protector is a recently introduced, improved version the LMA supreme - another second generation SAD. LMA supreme has been used in clinical practice for more than 10 years, however, tracheal intubation through the device was extremely difficult because of the small size of the breathing channel. The LMA Protector, has a larger breathing channel allowing the passage of an endotracheal tube. Compared to the I-gel, is has also got a larger gastric drainage tube. This allows easy suction in the event of regurgitation. Therefore, it appears to be superior to the I-gel in preventing the aspiration. But there are no studies comparing the ease of intubation through I-gel and LMA Protector

The aim of this study is to compare the ease of performing the fibreoptic guided tracheal intubation through these two devices. Our hypothesis is that intubation through the I-gel is easier and quicker.

ELIGIBILITY:
Inclusion Criteria:

• All patients aged above 18, presenting for elective surgical procedure, where a supraglottic airway device can be used and left in place throughout the duration of surgery and requiring tracheal intubation

Exclusion Criteria:

* Patients who are do not wish to take part
* Patients with class II obesity (BMI >40)
* Patients below 18 years of age
* American Society of Anaesthesiologists (ASA 3, 4 and 5)
* Patients with mouth opening of less than 3 cm
* Patients deemed to require awake intubation
* Surgery involving head and neck region
* Surgery requiring prone position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyprian Mendonca, Prof., Principal Investigator — University Hospitals Coventry & Warwickshire NHS Trust, Clifford Bridge Road, Coventry CV2 2DX
Locations (2):
- United Kingdom (2):
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands
  - Oxford University Hospitals, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Kleine-Brueggeney M, Theiler L, Urwyler N, Vogt A, Greif R. Randomized trial comparing the i-gel and Magill tracheal tube with the single-use ILMA and ILMA tracheal tube for fibreoptic-guided intubation in anaesthetized patients with a predicted difficult airway. Br J Anaesth. 2011 Aug;107(2):251-7. doi: 10.1093/bja/aer103. Epub 2011 Jun 7. PMID 21652616
- [Background] El-Ganzouri, A. R., Marzouk, S., Abdelalem, N., & Yousef, M. (2011). Blind versus fiberoptic laryngoscopic intubation through air Q laryngeal mask airway. Egyptian Journal of Anaesthesia, 27(4), 213-218.
- [Background] Taxak, S., Vashisht, K., Kaur, K. P., Ahlawat, G., & Bhardwaj, M. (2013). A study to evaluate fibreoptic-guided intubation through the i-gel. Southern African Journal of Anaesthesia and Analgesia, 19(2), 120-123.
- [Background] Samir, E. M., & Sakr, S. A. (2012). The air-Q as a conduit for fiberoptic aided tracheal intubation in adult patients undergoing cervical spine fixation: A prospective randomized study. Egyptian Journal of Anaesthesia, 28(2), 133-137.
- [Background] Jagannathan N, Sohn L, Ramsey M, Huang A, Sawardekar A, Sequera-Ramos L, Kromrey L, De Oliveira GS. A randomized comparison between the i-gel and the air-Q supraglottic airways when used by anesthesiology trainees as conduits for tracheal intubation in children. Can J Anaesth. 2015 Jun;62(6):587-94. doi: 10.1007/s12630-014-0304-9. Epub 2014 Dec 24. PMID 25537736
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Joffe AM, Liew EC, Galgon RE, Viernes D, Treggiari MM. The second-generation air-Q intubating laryngeal mask for airway maintenance during anaesthesia in adults: a report of the first 70 uses. Anaesth Intensive Care. 2011 Jan;39(1):40-5. doi: 10.1177/0310057X1103900106. PMID 21375088

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | I-gel | LMA Protector
Started | 90 | 90
Treated | 2 | 0
Failed | 0 | 4
Completed | 90 | 86
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I-gel | LMA Protector | Total
Number analyzed (Participants) | 90 | 86 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 55 | 112
  >=65 years | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (15) | 54.7 (17) | 55 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 51 | 51 | 102
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 90 | 86 | 176

OUTCOME MEASURES:

1. Primary Outcome: Total Intubation Time to Perform Fibreoptic Intubation
Description: Time form insertion of bronchoscope through the supraglottic airway device to obtaining the capnography trace
Time Frame: less than 3 minutes
Population: In 2 patients randomly allocated to the LMA Protector group due to the failure insertion of the LMA protector the i-gel was used instead. 2 patients randomised to the LMA protector group underwent direct laryngoscopy and tracheal intubation; one due to failed insertion of both devices and one due to the failed fibreopitc-guided tracheal intubation
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-gel | LMA Protector
Number analyzed (Participants) | 92 | 86
seconds | 54.3 (13.8) | 52.0 (13)

2. Secondary Outcome: SAD Insertion Time
Description: Time taken to insert the supra-glottic airway device measured from insertion into the mouth until the capnography trace is obtained
Time Frame: less than 1 minute
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-gel | LMA Protector
Number analyzed (Participants) | 92 | 86
seconds | 19.4 (5.6) | 25.4 (7.9)

3. Secondary Outcome: Number of Attempts at the SAD Placement
Description: Number of attempts taken to successfully place the supraglottic airway device in the oropharynx
Time Frame: less than 2 minutes
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants With Ease of Placement of the SAD
Description: The ease of placement of the SAD assessed by the investigator on a four point scale:
  1. - Easy
  2. - Moderate Difficulty 3- Severe Difficulty
  4 - Failure
Time Frame: less than 2 minutes
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | I-gel | LMA Protector
Number analyzed (Participants) | 92 | 86
participants
  Easy | 86 | 37
  Moderate Resistance | 6 | 44
  Severe Resistance | 0 | 5
  Failure | 0 | 0

5. Secondary Outcome: Number of Participants With First and Second Attempt at Tracheal Intubation
Description: Number of attempts at tracheal intubation. A new attempt is defined as re-insertion of the fibreoptic bronchoscope through the SAD.
Time Frame: less than 3 minutes
Population: IIn 2 patients randomly allocated to the LMA Protector group due to the failure insertion of the LMA protector the i-gel was used instead. 2 patients randomised to the LMA protector group underwent direct laryngoscopy and tracheal intubation; one due to failed insertion of both devices and one due to the failed fibreopitc-guided tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | I-gel | LMA Protector
Number analyzed (Participants) | 92 | 86
Participants
  First Attempt | 90 | 84
  Second Attempt | 2 | 2

6. Secondary Outcome: Number of Participants With Quality of the View of the Vocal Cords Seen Through the SAD
Description: The quality of the view of the vocal cords seen through the SAD. It will be assessed, according to the previously published system, as: grade I - full view of the vocal cord, II - partial view of the vocal cords including arytenoids, III - epiglottis only, IV - other (SAD cuff, pharynx, others)
Time Frame: less than 3 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | I-gel | LMA Protector
Number analyzed (Participants) | 92 | 86
Participants
  Grade 1 | 71 | 72
  Grade 2 | 20 | 14
  Grade 3 | 1 | 0

7. Secondary Outcome: Time to Carinal View
Description: The time from insertion of fibreoptic scope into the lumen of the SAD to the visualization of the carina.
Time Frame: less than 1 minute
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-gel | LMA Protector
Number analyzed (Participants) | 92 | 86
seconds | 23.4 (10) | 21.9 (8.3)

8. Secondary Outcome: Number of Participants With Type of Airway Maneuvers Performed During Tracheal Intubation,
Description: The number of tube rotations performed during tracheal intubation
Time Frame: less than 3 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | I-gel | LMA Protector
Number analyzed (Participants) | 92 | 86
Participants
  Tube impingement (Yes) | 38 | 23
  Tube impingement (No) | 54 | 63

ADVERSE EVENTS:
Time Frame: 1 year
Description: In two patients randomly allocated to the LMA protector group, due to failed insertion of LMA protector the I-GEL was used instead In two patients allocated to the LMA protector group, due to failed intubation direct laryngoscopy was performed.
  Therefore; the final number in I-GEL group is 92 and LMA Protector Group is 86(2 were allocated to I-GEL and 2 completely failed)
Arm/Group | I-gel | LMA Protector
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/86
Other Adverse Events (participants affected / at risk) | 0/92 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT03118596/Prot_SAP_000.pdf